CLINICAL TRIAL: NCT02058238
Title: ADDRESS - Multicenter, Partially-randomized Controlled Trial of Adult Deformity Robotic vs. Freehand Surgery to Correct Adult Spine Deformity
Brief Title: ADDRESS - Adult Deformity Robotic vs. Freehand Surgery to Correct Spinal Deformity
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Mazor Robotics (Industry)
Responsible Party: Sponsor
Other Study IDs: CLN105
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Scoliosis; Kyphosis; Kyphoscoliosis; Spinal Deformity; Spondylosis
Keywords: Robotic-guided spinal fusions; Scoliosis; Kyphoscoliosis; Spinal deformity; Spondylosis
MeSH Terms: conditions — Scoliosis; Kyphosis; Spondylosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Arm 1: Robotic-guided, Open approach: Adult patients (age> 21 years) undergoing long (>4 consecutive vertebrae) open instrumentation, correction and fusion surgery in the thoracic, lumbar or sacral spine for a kypho/scoliotic curve, sagittal or coronal imbalance or a combination of these.
- Arm 2: control-arm - non-robotic, open approach: Adult patients (age> 21 years) undergoing long (>4 consecutive vertebrae) open instrumentation, correction and fusion surgery in the thoracic, lumbar or sacral spine for a kypho/scoliotic curve, sagittal or coronal imbalance or a combination of these.
- Arm 3: robotic-guided, MIS approach: Adult patients (age> 21 years) undergoing long (>4 consecutive vertebrae) open instrumentation, correction and fusion surgery in the thoracic, lumbar or sacral spine for a kypho/scoliotic curve, sagittal or coronal imbalance or a combination of these.
- Arm 4: control-arm - freehand, MIS approach: Adult patients (age> 21 years) undergoing long (>4 consecutive vertebrae) open instrumentation, correction and fusion surgery in the thoracic, lumbar or sacral spine for a kypho/scoliotic curve, sagittal or coronal imbalance or a combination of these.

SUMMARY:
To quantify potential short- and long-term benefits of robotically-guided minimally invasive (MIS) or open-approach spine surgery in adult patients undergoing multi-level spinal instrumentation surgery, in comparison to image- or navigation-guided instrumentation in a matching cohort of control patients, performed using a freehand technique, both in MIS and open approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (age 21 years and older), undergoing long (5 consecutive vertebrae or more) spinal fusion surgery, between T1 to the sacrum.
2. Cases may include surgeries involving iliac screws (e.g., Galveston technique or S2AI screws) although these screws will not be included in the data analysis.
3. Cases may include augmented cases (when one or more of the screws are inserted into vertebrae after a vertebral augmentation procedure, such as kyphoplasty or vertebroplasty).
4. Patient capable of complying with study requirements
5. Signed informed consent by patient

Exclusion Criteria:

1. Infection or malignancy
2. Primary abnormalities of bones (e.g. osteogenesis imperfecta)
3. Primary muscle diseases, such as muscular dystrophy
4. Neurologic diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, cerebral palsy, spina bifida, or neurofibroma)
5. Spinal cord abnormalities with any neurologic symptoms or signs
6. Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia
7. Paraplegia
8. Patients who have participated in a research study involving an investigational product in the 12 weeks prior to surgery
9. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study.
10. Pregnancy
11. Patient cannot follow study protocol, for any reason
12. Patient cannot or will not sign informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age over 21 years) undergoing long (5 or more consecutive vertebrae) open or minimally invasive instrumentation, correction and fusion sugery in the thoracic, lumbar or sacral spine who have been found to have kypho/scoliotic curve, sagittal or coronal imbalance or a combination of these.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-10-03 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2015-03-01 (Actual)

PRIMARY OUTCOMES:
Incidence of surgical complications | 1 year
  New neural deficits, implant-related durotomy, infection requiring surgery, excessive blood loss
Intraoperative radiation exposure | Day of operation
  as measured by the C-arm, normalized per screw
Revision surgeries | 2 years
  All cause revisions, including medical and surgical complications.

SECONDARY OUTCOMES:
Deformity correction as measured on plain radiographs | Within 2 years from surgery
  Parameters of sagittal and coronal balance
Clinical outcome measures assessed using health-related quality of life questionnaires | up to 10 years post-operative
  Visual Analog Scale (VAS) back and leg, Oswestry Disability Index (ODI), SRS22 questionnaire, European Quality - 5 dimensions (EQ-5D-5L)
Pedicle screw instrumentation accuracy | Within 1 year of surgery
  Accuracy will be quantified in millimeters and scored using the Gertzbein Robbins classification, based on post-operative CTs that are clinically necessary for the management of the patient.
Length of convalescence | Within 2 years of surgery
  Length of stay at the hospital, destination at discharge, time to return to normal activities, time to return to work
Ratio of executed vs. planned screws | Day of surgery
  Number of screws planned to be robotically inserted but manually inserted instead, and cause.
Times of intra-operative stages | Day of surgery
  Instrumentation time per screw, total surgery time
Implant Failure | Within 1 year post-surgery
  The implant failure rate as measured within one year post-surgery
Number of Abandoned Screws | Day of surgery
  Number of screws intended to be instrumented with the robot and abandoned for cause.
Number of screws instrumented freehand | Day of surgery
  Number of screws planned to be instrumented robotically and instrumented freehand instead.
Clinical performance of instrumentation technique | Day of surgery
  Implant instrumentation time, length of surgery
Fusion rate/pseudoarthrosis | Within one year post-surgery
  Fusion/pseudoarthrosis as measured within one year of surgery
Neuromonitoring events | Day of surgery
  The number of clinically significant neuromonitoring events that may or may not lead to removal or reinstrumentation of the pedicle screw.

CONTACTS AND LOCATIONS:
Overall Officials: Doron Dinstein, MD, Study Director — Mazor Robotics
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Background] Hu X, Ohnmeiss DD, Lieberman IH. Use of an ultrasonic osteotome device in spine surgery: experience from the first 128 patients. Eur Spine J. 2013 Dec;22(12):2845-9. doi: 10.1007/s00586-013-2780-y. Epub 2013 Apr 16. PMID 23584231
- [Background] Devito DP, Kaplan L, Dietl R, Pfeiffer M, Horne D, Silberstein B, Hardenbrook M, Kiriyanthan G, Barzilay Y, Bruskin A, Sackerer D, Alexandrovsky V, Stuer C, Burger R, Maeurer J, Donald GD, Schoenmayr R, Friedlander A, Knoller N, Schmieder K, Pechlivanis I, Kim IS, Meyer B, Shoham M. Clinical acceptance and accuracy assessment of spinal implants guided with SpineAssist surgical robot: retrospective study. Spine (Phila Pa 1976). 2010 Nov 15;35(24):2109-15. doi: 10.1097/BRS.0b013e3181d323ab. PMID 21079498